CLINICAL TRIAL: NCT04510467
Title: Mental Health Consequences of COVID19 Infection in the French Rheumatic Musculoskeletal Diseases (RMD) Cohort
Brief Title: Mental Health Consequences of COVID19 Infection in the French RMD Cohort
Acronym: MentCovid19RMD
Status: Terminated | Type: Observational
Why Stopped: inclusion number not reached during the period
Sponsor: University Hospital, Lille (Other)
Collaborators: FAI²R (Auto-immune and auto-inflammatory rare diseases French network) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020_75; 2020-A02058-31 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-08-11; First posted 2020-08-12 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Covid19; Systemic Autoimmune Disease; Inflammatory Rheumatism; Auto Inflammatory Diseases
MeSH Terms: conditions — COVID-19; Rheumatic Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case group: RMD patients with COVID 19 infection
- control group: RMD patients without COVID 19 infection

SUMMARY:
this observational, cross-sectional, national, comparative study, including RMD patients followed in hospital centres of the FAI²R Rare Diseases Healthcare Pathway network and specialist private practitioners caring for patients suffering from inflammatory rheumatism, systemic autoimmune diseases and auto-inflammatory diseases. The objective of the study is to compare RMD patients with COVID 19 infection (cases) to RMD patients who have not had COVID 19 infection (controls) on their mental health.

ELIGIBILITY:
Inclusion Criteria:

Patient case:

* Patient with inflammatory rheumatism, systemic autoimmune or autoimmune disease
* With confirmed COVID-19 infection (at least one month prior to study inclusion)
* Study information given to the patient
* Patient affiliated to social security

Patient control:

* Patient with inflammatory rheumatism, systemic autoimmune disease or autoimmune disease.
* Not having had a confirmed COVID-19 infection
* Study information given to the patient
* Patient affiliated to social security

Exclusion Criteria:

* Opposition to participation in the study by the patient and/or his legal representative
* Adult patient not able to understand the implications and rules of the study
* Protected adults under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the French RMD covid19 cohort (ClinicalTrials.gov Identifier: NCT04353609) including patients from hospitals in the FAI²R Rare Diseases Healthcare Pathway network and specialist private practitioners (rheumatologists, internists with mixed hospital and private practice activities) caring for patients with inflammatory rheumatism, systemic autoimmune diseases and auto-inflammatory diseases.
Sampling Method: Probability Sample
Enrollment: 296 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Frequency of PTSD depending on whether or not autoimmune patients have experienced COVID | at one month following exposure to the traumatic factor (i.e. one month from COVID-19 infection

SECONDARY OUTCOMES:
Severity of PTSD depending on whether or not autoimmune patients have experienced COVID | at one month following exposure to the traumatic factor (i.e. one month from COVID-19 infection

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hachulla, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France